CLINICAL TRIAL: NCT02854878
Title: Treatment of Head Lice Infestation Using Novel Ultrasonic Comb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ParaSonic Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-001
Record Dates: First submitted 2016-07-26; First posted 2016-08-04 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Pediculus Capitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental)
  Interventions: Device: The Lucy ultrasonic comb models A and B combined with the LucyGel

INTERVENTIONS:
Device: The Lucy ultrasonic comb models A and B combined with the LucyGel

SUMMARY:
A pilot study to evaluate safety and efficacy of the Lucy combined with LucyGel in killing head lice and their eggs.

23 participants will be enrolled in this study. The first 12 will be combed with model A and the remaining 11 will be combed with model B

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* Age 6 years and older at the time of enrollment
* Must have an active head lice infestation of at least 10live head lice (found within 5 minutes of mechanic search).
* Hair must be at least 3 cm long.
* Written informed consent - by patient (if over 18 years of age), or by a parent (if patient is under 18 years of age).
* For females of childbearing potential, a statement declaring that she is not currently pregnant.

Exclusion Criteria:

* Used any chemical head lice treatment in the 7 days preceding the trial treatment
* Used antibiotics in the week preceding treatment
* Open wounds in the treatment area
* Skin irritation in the treatment area
* Individuals with skin/scalp condition at the treatment site which, in the opinion of the investigator, will interfere with treatment or evaluation
* Known allergies to any of the gel's components
* Participant that is already enrolled in another study
* Participant who can't be combed with fine Comb dense ASSY2000

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Adverse events of the device and treatment | up to three days
  measured by AE

SECONDARY OUTCOMES:
Mortality of up to 70% of the mature head lice 3 hours post treatment | 3 hours post treatment
Mortality of up to 50% of the head lice eggs 14 days post treatment. | 14 days post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Herzeliya medical center, Herzliya, Israel